CLINICAL TRIAL: NCT05336929
Title: Effect of Roy Adaptation Model on Metabolic Control in Adolescents With Type 1 Diabetes: Randomized Controlled Trial
Brief Title: Roy Adaptation Model in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Collaborators: Uludag University (Other)
Responsible Party: Principal Investigator, Gulsah Sunay Ertem, Msc, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Balıkesir University
Record Dates: First submitted 2022-03-23; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes; Adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education arm (n=30) (Experimental): Roy adaptation model-based training was given to the training arm.
  Interventions: Other: Roy adaptation model-based nursing education
- control arm (n=30) (No Intervention): Roy adaptation model-based training not given to the training arm

INTERVENTIONS:
Other: Roy adaptation model-based nursing education
  Arms: education arm (n=30)

SUMMARY:
The study was conducted to determine the effect of Roy adaptation model-based education on disease compliance and metabolic control in adolescents with Type 1 diabetes.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled study. A total of 60 adolescents, training (n=30) and control (n=30) that meet the research criteria were divided by random method. Pre-training data of the groups were collected using the "Sociodemographic Form", "Diabetes Information Evaluation Form" and "Roy Adaptation Model Interview Form" and HbA1c values were recorded. The training group was trained on the Roy Adaptation Model by a month break, in two sessions. After the training, the adolescents in the training group were given a curvature booklet based on the Roy Adaptation model. The control group was not intervened. After the training, the diabetes Information Assessment Form and the Roy Adaptation Model Discussion Form have applied to both groups again and the values of HbA1c were recorded.

ELIGIBILITY:
Inclusion criteria:

1. Having type 1 diabetes
2. Must be between the ages of 11-18
3. volunteering for research

Exclusion criteria

1. Presence of mental disability
2. To have received training on the content of the study

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c values | 3 month
  change from baseline in HbA1c value at 3 months

SECONDARY OUTCOMES:
Diabetes Knowledge Level | baseline and 2nd month
  change from baseline in diabetes knowledge level on the 32 points diabetes knowledge level form at month 2

OTHER OUTCOMES:
Roy Adaptation Model Interview results | baseline and 2nd month
  Change of adaptation behavior to illness consisting of 27 questions in 2 months

CONTACTS AND LOCATIONS:
Overall Officials: sibel ergün, Assoc. Dr., Principal Investigator — sibel.ergun@balikesir.edu.tr

IPD SHARING:
Plan to Share IPD: No